CLINICAL TRIAL: NCT00954616
Title: Inappropriate Medications and Alzheimer Disease: Prevalence and Associated Factors in Elderly Patients Treated With Anticholinesterase and/or Memantine. MIDA Study.
Brief Title: Inappropriate Medications Associated With Anticholinesterase and/or Memantine Treatment in the Elderly
Acronym: MIDA
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I07033
Record Dates: First submitted 2009-07-31; First posted 2009-08-07 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2009-08

CONDITIONS: Alzheimer's Disease
Keywords: Inappropriate Medications Associated; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In each of the 7 French areas that should be involved, patients aged 75 years and over from three different sectors will be included: the geriatric consultation unit (60%) and two kinds of nursing homes, private (20%) and state (10%). Outpatients will be included in chronological order; patients in nursing homes will be included at random. The patients and their families will be asked about the treatments received on the day of inclusion. The inclusion period will extend over a year. The investigating practitioners will be asked to fill in a questionnaire reporting the main clinical data, adverse effects occurrence, and information on the treatment given.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 years and over identified as having Alzheimer disease and who have been treated for more than 3 months with anticholinesterase and/or memantine

Exclusion Criteria:

* Patients with decompensated chronic condition or acute phase disease

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient of 75 and more years old affected by the Alzheimer's disease
Sampling Method: Probability Sample
Enrollment: 636 (Actual)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the prevalence of PIM use in patients aged 75 years and over treated with anticholinesterase and/or memantine | 2 years

SECONDARY OUTCOMES:
To identify factors associated with PIM use. To study the relationship between PIM exposure and adverse effects occurrence. | 2 years

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU Rouen, Rouen, Bois Guillaume
  - CHU Bordeaux, Pessac, Bordeaux
  - CH Le Mans, Le Mans, Le Mans Cedex 1
  - CHU Montpellier, Montpellier, Montpellier Cedex 5
  - APHP Charles Foix, Ivry-sur-Seine, Paris
  - CHU Saint Etienne, Saint-Etienne, Saint Etienne